CLINICAL TRIAL: NCT05284292
Title: GUARDIAN: The Social Robot Companion to Support Homecare Nurses
Acronym: GUARDIAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INRCA_001_2022
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Aging Problems; Caregiver
Keywords: Health informatics; Attitude to computers; Technology; Technological Innovations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): The Guardian platform consists of the robot Misty II, the Senior App and the Caregiver App will be tested by the elderly subjects together with their caregivers
  Interventions: Device: GUARDIAN platform

INTERVENTIONS:
Device: GUARDIAN platform — The enrolled elderly subjects and their caregivers will use at home the GUARDIAN platform consists of the Senior App, the Caregiver App and the Misty II robot.

SUMMARY:
The primary objective of this study is to verify the acceptability of the GUARDIAN system by the elderly, detected through the scale Unified Theory of Acceptance and Use of Technology (UTAUT). The GUARDIAN platform consists of two connected apps: one dedicated to the caregiver and one dedicated to the older people, plus a robot (Misty II). Misty II will live with the elderly, it will have the task of detecting his presence inside the house, reminding him of appointments, assisting him in his daily activities and diminishing the sense of loneliness. The application dedicated to the caregiver receives the data and self reports of the elderly from the robot, in order to constantly offer an updated picture of the condition of the elderly and to keep them informed about their condition and well-being.

DETAILED DESCRIPTION:
The primary objective of this study is to verify the acceptability of the GUARDIAN platform by the elderly, detected through the scale Unified Theory of Acceptance and Use of Technology (UTAUT). The aim of this project is to enable the older adult to live as long as possible at home, involving the informal caregiver, using the available technologies. The GUARDIAN platform consists of the Senior App, the Caregiver App and the Misty II robot. The Senior App is an easy-to-use application that will ask the elderly for health status, whether they have carried out their daily activities, if they have taken pre-establishable drugs and if they have eaten properly. The application will generate self-reports that will be transmitted to the app caregiver. The elderly can answer the questions via a tablet on the robot or by voice. The Caregiver App is the application intended for the caregiver, in which you can set up reminders for the elderly about meals or drugs, send communications and ask for reports on his health. This application will be used by both the informal caregiver and the formal caregiver (health care professional). It is the social robot that will complete the platform. Reminders will be sent via the robot and questions will be asked to the patient. The trial will consist of two phases involving, in each of the three participant countries (Italy, Nederlands and Switzerland), 4 seniors with their informal caregivers in the Alpha phase and 10 seniors with their informal caregivers in the following GUARDIAN trial. In both phases the presence of a formal caregiver is expected. In the Alpha phase 4 users and their caregivers will use a first version of the GUARDIAN platform, for three months. The results and feedback from the Alpha phase will give indications to improve and refine the platform.

The GUARDIAN trial involves the enrollment of 10 elderly people in each of the three participant countries (different from those recruited in the Alpha phase) and their respective informal caregivers. The evaluations will be carried out at baseline (T0) and then every month, for three months (T1, T2, T3).

ELIGIBILITY:
Inclusion Criteria:

* Cognitive integrity (Mini Mental State Examination >=24)
* Have an informal caregiver
* Healthy sight and hearing

Exclusion Criteria:

* Mini Mental State Examination < 24
* Lack of informal caregivers
* Sight and hearing not intact
* Lack of informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the acceptability of the GUARDIAN platform | change from baseline to 1, 2 and 3 months after intervention commencement
  Acceptability will be assessed using a 32-item questionnaire based on the unified theory of acceptance and use of technology (UTAUT) model. It's a standardized instrument for measuring the likelihood of success for new technology introductions and helps to understand the drivers of its acceptance.
  The questionnaire has 32 questions distributed in 4 key constructs: 1) performance expectancy, 2) effort expectancy, 3) social influence, and 4) facilitating conditions.
  Each question are based on a Likert-type 5-point scale ranging from 1 = strongly disagree to 5 = strongly agree. Increments are integers between 1 to 5.

SECONDARY OUTCOMES:
Care load of the informal caregiver | change from baseline to 1, 2 and 3 months after intervention commencement
  Zarit Burden Interview (Chattat R. et al. 2011)
Caregiver's Stress and Anxiety | change from baseline to 1, 2 and 3 months after intervention commencement
  The General Anxiety Disorder-7 (GAD-7) is used to measure the severity of anxiety. Score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively. When used as a screening tool, further evaluation is recommended when the score is 10 or greater.
Quality of life of the elderly | change from baseline to 1,2 and 3 months after intervention commencement
  The Euro QoL 5D-5L quality of life scale is a survey of perceived quality of life that consists of 5 domains: Mobility, self-care, usual activities, pain/discomfort and anxiety/depression; each domain is evaluated with an inverse Likert scale of 5 points where 1 indicates the absence of a problem and 5 the most extreme problem. It also consists of a subscale that evaluates the level of global health through a visual analog scale of 100 points. A unique health state is defined by combining 1 level from each of the 5 dimensions, this combination can be converted into a single index value by facilitating the calculation of quality-adjusted life years (QALYs).
Elderly person's perception of their health | change from baseline to 1, 2 and 3 months after intervention commencement
  SF-12 Health Survey (SF-12) is composed of 12 items that produce two measurements related to two different aspects of health: physical health and mental health

CONTACTS AND LOCATIONS:
Locations (3):
- Irccs Inrca, Ancona, Italy
- Hospital St Jansdal, Harderwijk, Netherlands
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

REFERENCES:
- [Derived] Margaritini A, Benadduci M, Amabili G, Bonfigli AR, Luzi R, Wac K, Nap HH, Maranesi E, Bevilacqua R. The social robot companion to support homecare nurses: The guardian study protocol. Contemp Clin Trials Commun. 2022 Oct 30;30:101024. doi: 10.1016/j.conctc.2022.101024. eCollection 2022 Dec. PMID 36340699